CLINICAL TRIAL: NCT03422510
Title: A Phase 2 Multicenter, Open Label, Randomized Study of Two Titration Regimens of Oral CXA-10 in Subjects With Primary Focal Segmental Glomerulosclerosis (FSGS)
Brief Title: FIRSTx - A Study of Oral CXA-10 in Primary Focal Segmental Glomerulosclerosis (FSGS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Complexa, Inc. (Industry)
Collaborators: Kidney Research Network, formerly NephCure Accelerating Cures Institute (Unknown); Medpace, Inc. (Industry); MicroConstants (Unknown); Arkana Labs (Unknown); NephCure Kidney International (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CXA-10-204
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Primary Focal Segmental Glomerulosclerosis
Keywords: FSGS; Kidney Disease; Proteinuria; Nephrotic Syndrome; FIRSTx; Nitro fatty acids; OA-NO2; 10-nitro oleic acid; Nitro oleic acid
MeSH Terms: conditions — Kidney Diseases; Proteinuria; Nephrotic Syndrome | interventions — CXA-10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Regimen 1 - CXA-10 75 mg (Experimental): Subjects in regimen 1 will start at 75 mg and may stay at 75 mg or increase to 150 mg. This treatment arm stays at 75 mg.
  Interventions: Drug: CXA-10
- Regimen 1 - CXA-10 150 mg (Experimental): Subjects in regimen 1 will start at 75 mg and may stay at 75 mg or increase to 150 mg. This treatment arm increases to 150 mg.
  Interventions: Drug: CXA-10
- Regimen 2 - CXA-10 150 mg (Experimental): Subjects in regimen 2 will start at 150 mg and may stay at 150 mg or increase to 300 mg. This treatment arm stays at 150 mg.
  Interventions: Drug: CXA-10
- Regimen 2 - CXA-10 300 mg (Experimental): Subjects in regimen 2 will start at 150 mg and may stay at 150 mg or increase to 300 mg. This treatment arm increases to 300 mg.
  Interventions: Drug: CXA-10

INTERVENTIONS:
Drug: CXA-10 — CXA-10 (10-nitro-9(E)-octadec-9-enoic acid) is a specific isomer of nitro-oleic acid (OA-NO2)

SUMMARY:
This is a multicenter, open label, randomized study investigating two dose titration regimens of CXA-10 in subjects at least 18 years of age with primary FSGS.

The study will be performed at approximately 25 study centers across the United States of America (USA). The recruitment period is anticipated to be up to approximately 16 months. Approximately 30 subjects will be randomized to ensure 26 subjects complete the study. An optional 9 month open label is available

DETAILED DESCRIPTION:
This is a multicenter, open label, randomized study investigating two dose titration regimens of CXA-10 in subjects at least 18 years of age with primary FSGS.

The study will be performed at approximately 25 study centers across the United States of America (USA). The recruitment period is anticipated to be up to approximately 16 months. Approximately 30 subjects will be randomized.

Study participation for each subject will last up to 5 months. The study will consist of a screening period not to exceed 30 days (1 month), 90-day (3 month) treatment period, and an approximate 28-day (1 month) follow-up period after the last dose of study medication. An optional 9 month open label is available.

ELIGIBILITY:
Inclusion Criteria:

1. have a diagnosis of primary FSGS confirmed with biopsy.
2. eGFR or 24-hour creatinine clearance ≥ 40 mL/min/1.73 m2 at Screening.
3. The subject has a Up/c ratio ≥ 2 g protein/g creatinine based on a 24 hour urine sample collected during Screening (one 24-hour collection between Day -30 and Day -8).
4. Unless there is an allergy or intolerance, subject must be on an ACEi and/or ARB regimen for a minimum of 4 weeks prior to their screening Up/c assessment. The ACEi and/or ARB regimen must be stable for a minimum of 2 weeks prior to screening Up/c assessment (and there are no plans to change the ACEi/ARB regimen over the course of the study).
5. If receiving simvastatin containing products: simvastatin (Zocor), Vytorin, or any other combination therapy containing simvastatin, the simvastatin dose should not exceed 20 mg/day.
6. Non-pregnant, non-lactating, female of childbearing potential who agrees to use a reliable method of contraception or female is of non-childbearing potential defined as surgically sterile (hysterectomy or bilateral tubal ligation) or post-menopausal.

Exclusion Criteria:

1. The subject has collapsing variant of FSGS on renal biopsy.
2. The subject has secondary FSGS.
3. The subject has diabetic nephropathy.
4. The subject has any other form of acquired (including biopsy proven obesity-induced FSGS) or hereditary glomerular nephropathy.
5. The subject has a prolonged QTcF interval.
6. The subject is hypertensive.
7. The subject has a history of clinically significant cardiovascular events, arrhythmias, recurrent fainting, palpitations, or family history of congenital prolonged QT syndromes or sudden unexpected death due to a cardiac reason.
8. The subject has any known bleeding disorders or significant active peptic ulceration in the opinion of the investigator that precludes enrollment into this study.
9. The subject has clinically significant anemia in the opinion of the investigator that precludes enrollment into this study.
10. The subject has a history of any primary malignancy, including a history of melanoma or suspicious undiagnosed skin lesions, with the exception of the following:

    1. Basal cell or squamous cell carcinomas of the skin,
    2. Cervical carcinoma in situ,
    3. Other malignancies curatively treated and with no evidence of disease for at least 5 years, or
    4. Prostate cancer which is not currently or expected, during the study, to undergo radiation therapy, chemotherapy, and/or surgical intervention, or to initiate hormonal treatment.
11. The subject has a history of organ transplantation.
12. The subject has a history of HIV.
13. At the time of Screening (Visit 1), the subject has any co-existing disease or condition.
14. Since the time of presentation of symptoms/diagnosis of FSGS: the subject has received systemic (oral or parenteral) high-dose, long-term corticosteroid therapy (prednisone or alternative glucocorticoid) to treat kidney disease
15. Subject has a history of immunosuppressant therapy (calcineurin inhibitors, rituximab, or other non-steroid immunosuppressants).
16. The subject has a history of herbal or natural medication use (including fish oil) within 2 weeks or 5 half-lives, whichever is longer, prior to Baseline
17. The subject is currently taking a drug that may affect the measurement of serum creatinine (e.g. cimetidine, Bactrim, Pyridium).
18. The subject is currently taking a newly prescribed drug or new prescription for an increased dose of an existing drug that is known to prolong the QTc interval and has been associated with Torsades de pointes (a list is provided in Appendix H). Note: Stable doses of these drugs are permitted (i.e., subject has received the same dose and regimen for at least 30 days prior to Screening [Visit 1] with no anticipated changes to the dose or regimen during the study).
19. The subject is currently taking endothelin receptor antagonists, dimethyl fumarate (Tecfidera™), orlistat, fibrates (fenofibrate, bezafibrate, gemfibrozil and ciprofibrate), niacin or lomatapide.
20. The subject has any of the following abnormal laboratories at Screening:

    1. Serologic evidence of HIV, hepatitis B, or hepatitis C based on HIV antibody, HBsAg, and HCV Ab,
    2. Absolute lymphocyte counts below the lower limit of normal of the reference range
    3. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 3.0X upper limit of normal (ULN), alkaline phosphatase > 2X ULN of liver origin, and total bilirubin >2X ULN. If all LFTs are within normal limits (WNL) and total bilirubin is elevated, examination of direct and indirect bilirubin may be conducted to evaluate for Rotor's/Gilbert's Syndrome. Subjects with Rotor's/Gilbert's Syndrome may be enrolled.
21. Female subject with a positive urine beta-human chorionic gonadotropin (β-hCG) test at Screening (Visit 1) (all females) or Baseline (Visit 2) (females of childbearing potential or with a history of bilateral tubal ligation in the absence of documented menopause).
22. The subject has received a live attenuated vaccine within 6 weeks prior to Baseline (Visit 2) or plans to receive a live attenuated vaccine during the study period.
23. The subject has a recent history (within one year prior to Screening [Visit 1]) of abusing alcohol or illicit drugs (including marijuana) or history of extensive illicit intravenous drug use.
24. Any other condition and/or situation that causes the Investigator to deem a subject unsuitable for the study (e.g., due to expected study medication non-compliance, inability to medically tolerate the study procedures, or a subject's unwillingness to comply with study-related procedures).
25. The subject has known hypersensitivity to CXA-10, its metabolites, or formulation excipients.
26. The subject has had treatment with any investigational drug or device within 30 days or 5 half-lives (whichever is longer) prior to Screening (Visit 1) (this includes investigational formulations of marketed products, inhaled and topical drugs), or plans to participate in another investigational drug or device study at any time during this study.
27. The subject weighs < 40 kg

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Reduction in proteinuria | 3 months
  overall reduction as measured by percent change from baseline

SECONDARY OUTCOMES:
The percent of subjects with of partial remission, modified partial remission, and complete remission | months 1, 2, 3
  percent change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Danoff, MD, Study Director — Complexa, Inc.
Locations (24):
- United States (24):
  - Alabama Neurology Consultants, Huntsville, Alabama
  - Cedars Sinai Medical Center, Los Angeles, California
  - Stanford University, Palo Alto, California
  - A.I. duPont Hospital for Children, Wilmington, Delaware
  - University of Miami, Miami, Florida
  - Nephrology Associates of Northern Illinois and Indiana (NANI), Chicago, Illinois
  - Northwest Louisiana Nephrology, Shreveport, Louisiana
  - Kidney Care and Transplant Services of New England, Springfield, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - St. Clair Nephrology Research, Roseville, Michigan
  - Clinical Research Consultants-KCMO, Kansas City, Missouri
  - Albert Einstein College of Medicine, Montefiore, The Bronx, New York
  - Metrolina Nephrology Associates, Charlotte, North Carolina
  - Levine Children's Hospital, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Northeast Clinical Research Center (NCRC), Bethlehem, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Nephrology Associates, Franklin, Tennessee
  - Texas Tech, Amarillo, Texas
  - Renal Disease Research Institute, DeSoto, Texas
  - El Paso Medical Research, El Paso, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - The Polyclinic, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Undecided